CLINICAL TRIAL: NCT02838225
Title: A Randomized, Phase II Study Comparing DA (Paclitaxel, Pirarubicin) With DAC ( Paclitaxel, Pirarubicin，Cyclophosphamide) as Postoperative Adjuvant Treatment for Early-stage Breast Cancer
Brief Title: DA Versus DAC as Postoperative Adjuvant Treatment for Early-stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiang SUN, Chief of Dept. Breast Surgery, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-BREAST-DA vs DAC
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

ARMS (2):
- DA (Experimental): docetaxel 75 mg/m², iv, day 1, doxorubicin 50 mg/m² or epirubicin 75mg/m², iv, day 1, every 3 weeks for 6 cycles
  Interventions: Drug: Docetaxel, Doxorubicin
- DAC (Active Comparator): docetaxel 75 mg/m², iv, day 1 doxorubicin 50 mg/m² or epirubicin 75mg/m², iv, day 1 Cyclophosphamide 500 mg/m², iv, day 1 every 3 weeks for 6 cycles
  Interventions: Drug: Docetaxel, Doxorubicin, Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel, Doxorubicin
  Arms: DA
Drug: Docetaxel, Doxorubicin, Cyclophosphamide
  Arms: DAC

SUMMARY:
Our study is a prospective, non-inferior, randomized phase II clinical trial, to compare the efficacy and safety profiles of DA versus DAC as adjuvant chemotherapy regimens for early-stage breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 and <= 70 years old.
* Performance status (Karnofsky index) >= 80.
* Histological diagnosis of invasive breast cancer (T1-T3,N0-1,M0). Time window between surgery and study randomization must be less than 60 days.
* Surgery must consist of mastectomy or conserving surgery with axillary lymph node dissection.
* Positive axillary lymph nodes defined as at least 1 out of 10 nodes with presence of disease. If sentinel node technique is used, sentinel node can be the only node affected.
* Status of hormone receptors, HER2 status, Ki-67 index and p53 in primary tumour. Results must be available before the end of adjuvant chemotherapy.
* Written informed consent. Patients are able to comply with treatment and study follow-up.
* Patients must not present evidence of metastatic disease.
* Normal electrocardiogram (EKG) in the 12 weeks prior to randomization. If needed, normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF).
* Laboratory results (within 14 days prior to randomization):

Hematology: neutrophils >= 2.0x10^9/l; platelets >= 100x10^9/l; hemoglobin >= 10 mg/dl; Hepatic function: total bilirubin <= 1 upper normal limit (UNL); SGOT and SGPT <= 2.5 UNL; alkaline phosphatase <= 2.5 UNL. If values of SGOT and SGPT > 1.5 UNL are associated to alkaline phosphatase > 2.5 UNL, patient is not eligible; Renal function: creatinine <= 175 mmol/l (2 mg/dl); creatinine clearance >= 60 ml/min.

* Complete stage workup during the 12 weeks prior to randomization (mammograms are allowed within a 20 week window). All patients must have a bilateral mammogram, thorax x-ray, abdominal echography and/or computed tomography (CT)-scan. If bone pain, and/or alkaline phosphatase elevation, a bone scintigraphy is mandatory. This test is recommended for all patients. Other tests: as clinically indicated.
* Negative pregnancy test done in the 14 prior days to randomization.

Exclusion Criteria:

* Prior systemic therapy for breast cancer.Or prior therapy with anthracyclines or taxanes (paclitaxel or docetaxel) for any malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments.
* Any T4 or N2-3 or M1 tumour.
* Pre-existing grade >= 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria version 2.0 [NCI CTC v-2.0]).
* Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled HA or high risk arrhythmias.
* History of neurological or psychiatric disorders, which could preclude the patients from free informed consent.
* Active uncontrolled infection.
* Active peptic ulcer; unstable diabetes mellitus.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumour curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Chronic treatment with corticosteroids.
* Contraindications for corticosteroid administration.
* Concomitant treatment with raloxifene, tamoxifen or other selective estrogen receptor modulators (SERMs), either for osteoporosis treatment or for prevention. These treatments must stop before randomisation.
* Concomitant treatment with other investigational products; participation in other clinical trials with a non-marketed drug in the 20 previous days before randomization.
* Concomitant treatment with another therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-01; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
Adverse event rate (CTCAE v. 3.0) | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years